CLINICAL TRIAL: NCT00998946
Title: A Phase 2, Single-arm, Open-label, Multi-center Study of Pralatrexate in Patients With Relapsed or Refractory B-cell Non-Hodgkin's Lymphoma
Brief Title: Study of Pralatrexate to Treat Participants With Relapsed or Refractory B-cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDX-015
Record Dates: First submitted 2009-10-19; First posted 2009-10-21 (Estimated); Results first posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Lymphoma, B-Cell
Keywords: Relapsed; Refractory; Non-Hodgkin's
MeSH Terms: conditions — Lymphoma, B-Cell; Recurrence | interventions — 10-propargyl-10-deazaaminopterin; Vitamin B 12; Folic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pralatrexate (Experimental): Participants received pralatrexate at an initial dose of 30 mg/m^2, as IV push over 30 seconds to 5 minutes via a patent free-flowing IV line containing normal saline on Days 1, 8 and 15 of a 4-week cycle (weekly for 3 weeks with 1 week of rest) until criteria for discontinuation per protocol were met. The initial dose of 30 mg/m^2 may be reduced to 20 mg/m^2 weekly, permitted per protocol defined criteria. If pralatrexate 20 mg/m^2/week was not tolerated, pralatrexate had to be discontinued. Dose re-escalation was not allowed once dose reduction was done.
  Participants had dietary supplement of vitamin B12 and folic acid along with pralatrexate. Vitamin B12, given as 1mg IM, within 10 weeks of start of pralatrexate dosing, every 8-10 weeks throughout the study and for at least 30 days post last dose of pralatrexate. Folic acid was given 1mg daily, orally, for at least 7 days prior to start of pralatrexate, throughout the study and for at least 30 days post last dose of pralatrexate.
  Interventions: Drug: Pralatrexate; Dietary Supplement: Vitamin B12; Dietary Supplement: Folic Acid

INTERVENTIONS:
Drug: Pralatrexate — Pralatrexate injection administered as intravenous (IV) push
  Other Names: FOLOTYN; PDX; (RS)-10-propargyl-10-deazaaminopterin
Dietary Supplement: Vitamin B12 — 1 mg intramuscular (IM) injection
  Other Names: Cyanocobalamin
Dietary Supplement: Folic Acid — Oral 1 mg tablet
  Other Names: Vitamin B9; Folate; Folacin

SUMMARY:
The purpose of this study is to determine whether pralatrexate, given with vitamin B12 and folic acid, is effective in the treatment of relapsed or refractory B-cell Non-Hodgkin's lymphoma (NHL). The study will also investigate the safety of pralatrexate with vitamin B12 and folic acid in this participant population. Additionally, this study includes the collection of blood samples to investigate the pharmacokinetics (PK) of pralatrexate in this participant population (PK is the activity of a drug in the body over a period of time, including how the drug is absorbed, distributed in the body, localized in the tissues, and excreted from the body).

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically confirmed, measurable (lesion or node =2 cm by CT [at least 1 cm if by spiral CT]) B-cell Non-Hodgkin's Lymphoma, using the Revised European American Lymphoma (REAL) World Health Organization (WHO) disease classification
* Progressive or persistent disease after ≥ 1 prior treatment(s)
* Recovered from toxic effects of prior treatment
* At least 4 weeks since most recent cytotoxic therapy
* Easter Cooperative Oncology Group (ECOG) performance status ≤ 2
* Adequate blood, liver, and kidney functions as defined by laboratory levels
* 1.0 mg/day orally of folic acid for at least 7 days prior & 1 mg intramuscular of vitamin B12 within 10 weeks of the planned start of pralatrexate
* Females of childbearing potential must agree to use medically acceptable birth control from start of pralatrexate until at least 30 days after the last administration of pralatrexate and must have a negative serum pregnancy test within 14 days prior to the first day of study treatment
* Males who are not surgically sterile must agree to use medically acceptable birth control from start of pralatrexate until at least 90 days after the last administration of pralatrexate
* Available for repeat dosing and follow-up
* Able to give written informed consent

Exclusion Criteria:

* Relapsed participants with diffuse large B-cell lymphoma (DLBCL) who are candidates for high-dose therapy and autologous stem cell transplantation (SCT) and for whom high-dose therapy and autologous SCT is a standard curative option
* Active concurrent malignancy (except non-melanoma skin cancer or carcinoma in situ of the cervix). If there is a history of prior malignancies other than those exceptions listed above, the participant must be disease-free for ≥ 5 years. Participants with other prior malignancies < 5 years before study entry may still be enrolled if they have received treatment resulting in complete resolution of the cancer and currently have no clinical, radiologic, or laboratory evidence of active or recurrent disease
* Congestive heart failure Class III/IV according to the New York Heart Association Functional Classification
* Uncontrolled hypertension
* Known human immunodeficiency virus (HIV)-positive diagnosis
* Symptomatic central nervous system (CNS) metastases or lesions for which treatment is required. Participants who received prophylactic CNS treatment are eligible.
* Participants who have undergone an allogeneic SCT
* Participants who have relapsed < 100 days from the time of an autologous SCT
* Participants with disease refractory to peripheral blood SCT or who have relapsed < 100 days from the time of transplant
* Active uncontrolled infection, underlying medical condition, or other serious illness that would impair the ability of the participant to receive protocol treatment.
* Major surgery within 14 days of enrollment
* Receipt of any conventional chemotherapy or radiation therapy (encompassing a substantial [> 10%] amount of bone marrow) within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to study treatment or planned use during the course of the study
* Receipt of systemic corticosteroids within 1 week of study treatment, unless participant has been taking a continuous dose of no more than 10 mg/day of prednisone or its equivalent for at least 1 month
* Use of any investigational drugs, biologics, or devices within 4 weeks prior to study treatment or planned use during the course of the study
* Previous exposure to pralatrexate
* Females who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Kootenai Cancer Center, Post Falls, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - Owsley Brown Frazier Cancer Center, Louisville, Kentucky
  - Overton Brooks VA Medical Center, Shreveport, Louisiana
  - Frontier Cancer Center and Blood Institute, Billings, Montana
  - New York University Hospital, New York, New York
  - Providence Cancer Center, Portland, Oregon
  - The West Clinic (ACORN), Memphis, Tennessee
  - Gundersen Lutheran, La Crosse, Wisconsin
  - University of Wisconsin, Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pralatrexate
Started | 29
Safety Population | 27 (Safety population included all participants who received at least 1 dose of the study drug.)
Completed | 20
Not Completed | 9
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1
Not completed — Death | 2
Not completed — Reason Unspecified | 3
Not completed — Enrolled but not Dosed | 2

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who received at least 1 dose of the study drug.
Arm/Group | Pralatrexate
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (14.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Objective response rate was defined as the percentage of participants with a complete response (CR) or a partial response (PR). Tumor response was evaluated on the basis of clinical and radiological criteria, assessed according to International Workshop Criteria (IWC) with or without positron emission tomography (PET) scans. Per IWC criteria CR is defined as complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease-related symptoms if present before therapy, and normalization of those biochemical abnormalities definitely assignable to non-Hodgkin's lymphoma (NHL) and PR is defined as >= 50% decrease in sum of the product of the perpendicular diameters (SPD) of the six largest dominant nodes or nodal masses and no increase in size of other nodes, liver or spleen.
Time Frame: Up to 24 months
Population: Efficacy Evaluable Population included participants who received at least 1 dose of protocol specified treatment and had measurable disease at baseline to be considered evaluable.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pralatrexate
Number analyzed (Participants) | 27
percentage of participants | 4 [0 to 19]

2. Secondary Outcome: Duration of Response (DOR)
Description: The Duration of Response was defined as the time (in months) from the date the measurement criteria were first met for CR or PR (whichever status was recorded first) until the first subsequent date that relapse or progression was documented. It was assessed according to IWC with or without PET, subject to its availability. Per IWC, progression was defined as a ≥50% increase from the nadir in the individual sum of the products of the diameters of any index lesion; the reappearance of pathology, enlargement of liver/spleen, or unequivocal progression of non-measurable disease or appearance of any new lesions.
Time Frame: Up to 24 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pralatrexate
Number analyzed (Participants) | 27
months | NA [NA to NA] — Median, upper limit and lower limit of 95% confidence interval (CI) was not estimable due to insufficient number of participants with event.

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival (PFS) was the duration of time (in months) from first administration of study treatment to date of first documented progression or death from any cause. It was based on tumor assessments made according to the IWC with or without PET scans, subject to their availability. Per IWC, progression was defined as a ≥50% increase from the nadir in the individual sum of the products of the diameters of any index lesion; the reappearance of pathology, enlargement of liver/spleen, or unequivocal progression of non-measurable disease or appearance of any new lesions.
Time Frame: Up to 24 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pralatrexate
Number analyzed (Participants) | 27
months | 3.6 [1.9 to 3.7]

4. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival was the time (in months) from first administration of study treatment until the date of death.
Time Frame: Up to 24 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pralatrexate
Number analyzed (Participants) | 27
months | NA [7.4 to NA] — Median and upper limit of 95% CI was not estimable due to insufficient number of participants with event.

ADVERSE EVENTS:
Time Frame: Up to 24 months
Description: Safety Population included all participants who received at least 1 dose of study drug.
Arm/Group | Pralatrexate
All-Cause Mortality (participants affected / at risk) | 11/27
Serious Adverse Events (participants affected / at risk) | 11/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pralatrexate (N=27)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Neutopenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac Failure Congestive (Cardiac disorders) | 1
Ear Pain (Ear and labyrinth disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 5
Pyrexia (General disorders) | 2
Catheter Related Infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Failure To Thrive (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Sinus Headache (Nervous system disorders) | 1
Mental Status Changes (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Laryngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pralatrexate (N=27)
Neutropenia (Blood and lymphatic system disorders) | 7
Atrial fibrillation (Cardiac disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 11
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 13
Sinus tachycardia (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Dry eye (Eye disorders) | 2
Vision blurred (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 6
Abdominal tenderness (Gastrointestinal disorders) | 1
Consitpation (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 7
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Gingival pain (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 12
Odynophagia (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Oral discomfort (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 2
Proctitis (Gastrointestinal disorders) | 1
Saliva altered (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 16
Vomiting (Gastrointestinal disorders) | 6
Asthenia (General disorders) | 2
Chest pain (General disorders) | 1
Chills (General disorders) | 4
Early satiety (General disorders) | 1
Fatigue (General disorders) | 21
Gait disturbance (General disorders) | 1
Mucosal inflammation (General disorders) | 3
Oedema peripheral (General disorders) | 6
Pain (General disorders) | 3
Pyrexia (General disorders) | 7
Seasonal allergy (Immune system disorders) | 1
Bacteraemia (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 3
Catheter related infection (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Tonsillitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Viral rhinitis (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Open wound (Injury, poisoning and procedural complications) | 2
Radius fracture (Injury, poisoning and procedural complications) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 3
Blood urea increased (Investigations) | 2
Haemoglobin decreased (Investigations) | 1
International normalised ratio increased (Investigations) | 1
Neutrophil count (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count (Investigations) | 2
Urine output decreased (Investigations) | 1
Weight decreased (Investigations) | 3
White blood cell count (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 4
Decreased appetite (Metabolism and nutrition disorders) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Fluid overload (Metabolism and nutrition disorders) | 1
Fluid retention (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 3
Hyponatraemia (Metabolism and nutrition disorders) | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Aphonia (Nervous system disorders) | 1
Burning sensation (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Lethargy (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Sinus headache (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Insomina (Psychiatric disorders) | 2
Dysuria (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 3
Nephrolithiasis (Renal and urinary disorders) | 1
Oliguria (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 2
Urinary tract pain (Renal and urinary disorders) | 1
Vaginal discharge (Reproductive system and breast disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 2
Petechiae (Skin and subcutaneous tissue disorders) | 1
Photodermatosis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 2
Hypotension (Vascular disorders) | 2
Orthostatic hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No